CLINICAL TRIAL: NCT01469910
Title: Safety, Tolerability, and Pharmacokinetics of Single Ascending Doses of Simotinib Hydrochloride in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIM-101
Record Dates: First submitted 2011-11-07; First posted 2011-11-10 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simotinib (Experimental)
  Interventions: Drug: Simotinib Hydrochloride
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Simotinib Hydrochloride — Single ascending doses: 25 mg、50 mg、100 mg、150 mg、225 mg、300 mg、400 mg、500 mg、600 mg、750 mg
  Arms: Simotinib
Drug: Placebo — Single ascending doses: 150 mg、225 mg、300 mg、400 mg、500 mg、600 mg、750 mg
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and pharmacokinetics of single ascending doses of Simotinib Hydrochloride in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy , male or female subjects
* Age of 18 to 45 years
* Body Mass Index (BMI) of 19 to 24 kg/m2; and a total body weight > 50 kg for male, > 45 kg for female
* Written informed consent signed and dated by the subject
* Subjects who are willing and able to comply with study procedures

Exclusion Criteria:

* Any clinically significant disease or surgery within 4 weeks prior to the beginning of the study
* Known hypersensitivity to the study drug or similar drugs
* History of any serious disease, including but not limited to circulatory system, endocrine system, central nervous system, hematology, immunology, metabolic diseases and psychiatric disorders
* History of gastrointestinal, hepatic, and renal diseases, affecting drug absorption and metabolism
* Any clinically significant abnormal clinical laboratory tests
* Abnormal ECG or vital signs
* A positive test for HIV antibody
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result
* History of alcohol consumption within six months of the study defined as: an average weekly intake of > 14 units
* History of regular tobacco use or nicotine containing products within three months prior to screening
* Consumption of too much tea or coffee (> 8 cups/day)
* Use of any drug, which inhibits or induces hepatic drug metabolism, within 30 days prior to the beginning of the study
* Use of any drug within 14 days prior to the beginning of the study
* Participate in other clinical trials within 30 days prior to the beginning of the study
* Blood donation within 30 days of dosing
* All female subjects must not be of child-bearing potential
* Pregnant or lactating women

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2011-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
The incidence and severity of adverse events | within 7 days following administration of study drug

SECONDARY OUTCOMES:
The maximum plasma concentration (Cmax) | 0.5 h, 1 h, 2 h, 3 h, 4 h, 5 h, 6 h, 8 h, 10 h, 12 h, 16h, 24 h, 36 h, 48 h
The time to Cmax (tmax) | 0.5 h, 1 h, 2 h, 3 h, 4 h, 5 h, 6 h, 8 h, 10 h, 12 h, 16h, 24 h, 36 h, 48 h
Area under the plasma concentration-time curve (AUC) | 0.5 h, 1 h, 2 h, 3 h, 4 h, 5 h, 6 h, 8 h, 10 h, 12 h, 16h, 24 h, 36 h, 48 h
The Terminal half-life (t1/2) | 0.5 h, 1 h, 2 h, 3 h, 4 h, 5 h, 6 h, 8 h, 10 h, 12 h, 16h, 24 h, 36 h, 48 h

CONTACTS AND LOCATIONS:
Overall Officials: Zeneng Cheng, MD, Principal Investigator — The Third Xiangya Hospital of Central South University
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China